CLINICAL TRIAL: NCT04142424
Title: A Phase I, Randomized, Single-blind, Placebo-controlled Study to Assess the Safety, Tolerability and Pharmacokinetics of AZD2693 Following Single Ascending Dose Administration in Male and Female Subjects of Non-childbearing Potential in Overweight But Otherwise Healthy Subjects, and Healthy Chinese and Japanese Subjects
Brief Title: A Study to Understand the Safety, Tolerability, and Activity of Drug in Body Over a Period of Time of AZD2693, in Subjects of Non-Childbearing Potential in Overweight But Otherwise Healthy Subjects, and Healthy Chinese and Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D7830C00001
Record Dates: First submitted 2019-10-22; First posted 2019-10-29 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Metabolic Disorders; Non-alcoholic Steatohepatitis
Keywords: Single-ascending-dose; First-in-human; Chinese; Japanese; Dyslipidemia; Type II diabetes mellitus; Non-alcoholic fatty liver disease
MeSH Terms: conditions — Metabolic Diseases; Non-alcoholic Fatty Liver Disease; Dyslipidemias; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Subjects in this study will be categorized as follows:
  1. Overweight/mildly obese, but otherwise healthy subjects: There will be 6 cohorts, with 8 subjects in each cohort.
  2. Japanese and Chinese subjects: There will be 2 cohorts for Japanese subjects, and one cohort for Chinese subjects, with 8 subjects in each cohort.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Cohort 1 healthy subjects: AZD2693 Dose 1 (Experimental): Subjects will receive a subcutaneous (SC) injection of single dose 1 of AZD2693 or placebo matched to AZD2693 on Day 1.
  Interventions: Drug: AZD2693; Drug: Placebo
- Cohort 2 healthy subjects: AZD2693 Dose 2 (Experimental): Subjects will receive a SC injection of single dose 2 of AZD2693 or placebo matched to AZD2693 on Day 1.
  Interventions: Drug: AZD2693; Drug: Placebo
- Cohort 3 healthy subjects: AZD2693 Dose 3 (Experimental): Subjects will receive a SC injection of single dose 3 of AZD2693 or placebo matched to AZD2693 on Day 1.
  Interventions: Drug: AZD2693; Drug: Placebo
- Cohort 4 healthy subjects: AZD2693 Dose 4 (Experimental): Subjects will receive a SC injection of single dose 4 of AZD2693 or placebo matched to AZD2693 on Day 1.
  Interventions: Drug: AZD2693; Drug: Placebo
- Cohort 5 healthy subjects: AZD2693 Dose 5 (Experimental): Subjects will receive a SC injection of single dose 5 of AZD2693 or placebo matched to AZD2693 on Day 1.
  Interventions: Drug: AZD2693; Drug: Placebo
- Cohort 6 healthy subjects: AZD2693 Dose 6 (Experimental): Subjects will receive a SC injection of single dose 6 of AZD2693 or placebo matched to AZD2693 on Day 1.
  Interventions: Drug: AZD2693; Drug: Placebo
- Cohort 7 healthy Japanese subjects: AZD2693 Dose 7 (Experimental): Subjects will receive a SC injection of single dose 7 of AZD2693 or placebo matched to AZD2693 on Day 1.
  Interventions: Drug: AZD2693; Drug: Placebo
- Cohort 8 healthy Japanese subjects: AZD2693 Dose 8 (Experimental): Subjects will receive a SC injection of single dose 8 of AZD2693 or placebo matched to AZD2693 on Day 1.
  Interventions: Drug: AZD2693; Drug: Placebo
- Cohort 9 healthy Chinese subjects: AZD2693 Dose 9 (Experimental): Subjects will receive a SC injection of single dose 9 of AZD2693 or placebo matched to AZD2693 on Day 1.
  Interventions: Drug: AZD2693; Drug: Placebo

INTERVENTIONS:
Drug: AZD2693 — Subjects will receive SC injection of AZD2693 as per the arms they are randomized.
Drug: Placebo — Subjects will receive SC injection of placebo matched to AZD2693, as per the arms they are randomized.

SUMMARY:
This Phase 1, first-in-human (FiH), single-ascending-dose (SAD) study, will assess the safety and tolerability and characterize the pharmacokinetics (PK) of AZD2693, following subcutaneous (SC) SAD administration of AZD2693 in male and female subjects of non-childbearing potential in overweight but otherwise healthy subjects, and healthy Chinese and Japanese subjects.

DETAILED DESCRIPTION:
This is a single center study, and approximately 64 overweight/mildly obese but otherwise healthy male and female subjects, and up to 16 healthy Japanese subjects and 8 healthy Chinese (all of non-childbearing potential) will be enrolled into this study.

Study will consist of following planned cohorts:

Eligible healthy subjects will be divided in 6 cohorts, each consisting of 8 subjects, within each cohort, 6 subjects will receive AZD2693 at dose level 1 and 2 subjects will receive placebo. Dosing for each ascending dose cohort will proceed with 2 subjects in a sentinel cohort, such that 1 subject will be randomized to receive placebo and 1 subject will be randomized to receive AZD2693.

Eligible healthy Japanese and Chinese subjects will be divided as two cohorts of Japanese subjects, and one cohort of Chinese subjects. Each cohort will consist of 8 subjects. Within each cohort, 6 subjects will receive AZD2693 and 2 subjects will receive placebo.

Depending on emerging data, up to 2 additional cohorts may be added to test additional dose levels based on Sponsor's decision.

Full study will comprise of following periods:

1. Screening period of maximum 28 days.
2. A Dosing Session during which subjects will be resident at the Clinical Unit from the day before investigational medicinal product (IMP) administration (Day -1) until at least 3 days after IMP administration with discharge on Day 4.
3. A Follow-Up Period of 16 weeks that will consist of 9 Follow-Up Visits, for which the subjects will return to the Clinical Unit at 1, 2, 4, 6, 8, 10, 12, 14, and 16 weeks post dose.

ELIGIBILITY:
Inclusion Criteria:

• Females must have a negative pregnancy test at the Screening Visit and on admission to the Clinical Unit, must not be lactating and must be of non-child-bearing potential, confirmed at the Screening Visit by fulfilling one of the following criteria: A. Postmenopausal defined as amenorrhea for at least 12 months or more following cessation of all exogenous hormonal treatments and follicle-stimulating hormone levels in the postmenopausal range B. Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation

* Have a body mass index between 25 and 32 kg/m^2 for healthy subjects, or between 18 and 32 kg/m^2 for healthy Japanese and Chinese subjects, and weigh at least 60 kg (or 50 kg for healthy Japanese and Chinese subjects)
* Willing to participate in mandatory retrospective genotyping analysis for PNPLA3 1148M and the provision of blood and buccal swab samples for this analysis
* Willing and able to comply with all required study procedures

Applicable to Japanese and Chinese subjects only:

* A Japanese subject is defined as having both parents and 4 grandparents who are ethnically Japanese. This includes second and third generation Japanese whose parents or grandparents are living in a country other than Japan
* A Chinese subject is defined as having both parents and 4 grandparents who are ethnically Chinese. This includes second and third generation Chinese whose parents or grandparents are living in a country other than China

Exclusion Criteria:

* History of any clinically important disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study
* History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs
* Any clinically important illness, medical/surgical procedure or trauma within 4 weeks of the first administration of IMP
* Any clinically significant cardiovascular event within the last 6 months prior to the Screening Visit
* Any laboratory values with the following deviations at Screening or Day -1:

  1. Alanine aminotransferase > upper limit of normal (ULN)
  2. Aspartate aminotransferase > ULN
  3. Creatinine > ULN
  4. White blood cell count < lower limit of normal (LLN)
  5. Hemoglobin < LLN
  6. Platelet count < LLN
  7. Activated partial thrombin time > ULN and prothrombin time > ULN
  8. Estimated glomerular filtration rate (eGFR) < 90 mL/min/1.73m^2 calculated using Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) and applying the standard correction factor for African Americans to the CKD-EPI by multiplying the GFR estimate by 1.159; (eGFR < 60 mL/min/1.73m^2 for healthy Japanese and Chinese subjects) and confirmed
  9. Urinary albumin-to-creatinine ratio > 3 mg/μmol (30 mg/g)
* Any other clinically important abnormalities in clinical chemistry, hematology or urinalysis results, than those described under previous exclusion criterion above, as judged by the Investigator at Screening or Day -1
* Any positive result on Screening for serum hepatitis B surface antigen, hepatitis C antibody and human immunodeficiency virus
* Abnormal vital signs, after 10 minutes supine rest, defined as any of the following at Screening or Day -1:
* Systolic BP < 90 mmHg or > 140 mmHg
* Diastolic blood pressure (BP) < 50 mmHg or > 90 mmHg
* HR < 45 or > 90 bpm
* Any clinically important abnormalities in rhythm, conduction or morphology of the resting electrocardiogram (ECG) and any clinically important abnormalities in the 12-lead ECG as considered by the Investigator that may interfere with the interpretation of QTc interval changes, including abnormal ST-T-wave morphology, particularly in the protocol defined primary lead or left ventricular hypertrophy at Screening or Day -1:
* Prolonged QTcF > 450 ms
* Shortened QTcF < 340 ms
* Family history of long QT syndrome
* PR (PQ) interval shortening < 120 ms (PR > 110 ms but < 120 ms is acceptable if there is no evidence of ventricular pre-excitation)
* PR (PQ) interval prolongation intermittent second (Wenckebach block while asleep is not exclusive) or third degree atrioventricular (AV) block, or AV dissociation
* Persistent or intermittent complete bundle branch block, incomplete bundle branch block, or intraventricular conduction delay with QRS > 110 ms Subjects with QRS > 110 ms but < 115 ms are acceptable if there is no evidence of e.g. ventricular hypertrophy or pre-excitation
* Known or suspected history of drug abuse as judged by the Investigator
* Smokers with > 10 cigarettes/day and unable to comply with the nicotine restrictions during the study
* History of alcohol abuse or excessive intake of alcohol. Definition of excessive intake: an average weekly intake of >21 drinks/week for men or >14 drinks/week for women. One drink is equivalent to (14 g alcohol)
* Positive screen for drugs of abuse at Screening or admission to the Clinical Unit or positive screen for alcohol on admission to the Clinical Unit prior to the first administration of the IMP
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the Investigator or history of hypersensitivity to drugs with a similar chemical structure or class to AZD2693
* Excessive intake of caffeine-containing drinks or food (e.g., coffee, tea, chocolate, Red Bull®-like drinks) as judged by the Investigator
* Use of any prescribed or nonprescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, mega-dose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks prior to the first administration of IMP or longer if the medication has a long half-life
* Plasma donation within one month of the Screening Visit or any blood donation/blood loss > 500 mL during the 3 months prior to the Screening Visit
* Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 30 days of last follow-up to first administration of IMP or, if known, 5 half-lives from last dose to first administration of IMP, whichever is the longest
* Blood dyscrasias with increased risk of bleeding including Idiopathic Thrombocytopenic Purpura and Thrombotic Thrombocytopenic Purpura or symptoms of increased risk of bleeding (frequent bleeding gums or nose bleeds)
* Involvement of any AstraZeneca or Clinical Unit employee or their close relatives
* Judgment by the Investigator that the subject should not participate in the study if they have any ongoing or recent (i.e., during the Screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions and requirements
* Subjects who are vegans or have medical dietary restrictions, or who are not willing to comply with the dietary requirements in the study as judged by the Investigator
* Subjects who cannot communicate reliably with the Investigator
* Vulnerable subjects, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order
* Previous bone marrow transplant
* Non-leukocyte depleted whole blood transfusion within 120 days of the date of the genotyping sample collection
* Males who are unwilling to use an acceptable method of birth control
* Subjects with a significant Coronavirus disease (COVID-19) illness within 6 months of enrollment:

a Subjects with diagnosis of COVID-19 pneumonia based on radiological assessment b Subjects with diagnosis of COVID-19 with significant findings from pulmonary imaging tests c Subjects with diagnosis of COVID-19 requiring hospitalization and/or oxygen supplementation therapy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2021-11-12 (Actual); Study Completion 2021-11-12 (Actual)

PRIMARY OUTCOMES:
Number of subjects experiencing adverse events and serious adverse events | From baseline (Day 1) until Day 112 (Week 16, Final follow-up)
  To investigate the safety and tolerability of SC administration of SAD of AZD2693

SECONDARY OUTCOMES:
Area under the concentration-time curve from time zero extrapolated to infinity (AUC) | At Day 1 pre-dose, 0.25 hours [h], 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 5h, 6h, 8h, 12h, 24h, 36h, 48h and 72h post-dose and 1, 2, 4, 8, 12 and 16 weeks post-dose
  To characterize the PK of AZD2693 following SC administration of SAD of AZD2693
Area under the plasma concentration-time curve from time zero to 48 hours after dosing [AUC(0-48h)] | At Day 1 pre-dose, 0.25h, 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 5h, 6h, 8h, 12h, 24h, 36h, 48h and 72h post-dose and 1, 2, 4, 8, 12 and 16 weeks post-dose
  To characterize the PK of AZD2693 following SC administration of SAD of AZD2693
Area under the plasma concentration-time curve from time zero to time of last quantifiable analyte concentration divided by the dose administered (AUClast/D) | At Day 1 pre-dose, 0.25h, 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 5h, 6h, 8h, 12h, 24h, 36h, 48h and 72h post-dose and 1, 2, 4, 8, 12 and 16 weeks post-dose
  To characterize the PK of AZD2693 following SC administration of SAD of AZD2693
Area under the plasma concentration-curve from time zero to the time of last quantifiable analyte concentration (AUClast) | At Day 1 pre-dose, 0.25h, 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 5h, 6h, 8h, 12h, 24h, 36h, 48h and 72h post-dose and 1, 2, 4, 8, 12 and 16 weeks post-dose
  To characterize the PK of AZD2693 following SC administration of SAD of AZD2693
Area under the plasma concentration-time curve from time zero extrapolated to infinity divided by the dose administered (AUC/D) | At Day 1 pre-dose, 0.25h, 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 5h, 6h, 8h, 12h, 24h, 36h, 48h and 72h post-dose and 1, 2, 4, 8, 12 and 16 weeks post-dose
  To characterize the PK of AZD2693 following SC administration of SAD of AZD2693
Maximum observed plasma drug concentration (Cmax) of AZD2693 | At Day 1 pre-dose, 0.25h, 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 5h, 6h, 8h, 12h, 24h, 36h, 48h and 72h post-dose and 1, 2, 4, 8, 12 and 16 weeks post-dose
  To characterize the PK of AZD2693 following SC administration of SAD of AZD2693
Observed maximum plasma concentration divided by the dose administered (Cmax/D) | At Day 1 pre-dose, 0.25h, 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 5h, 6h, 8h, 12h, 24h, 36h, 48h and 72h post-dose and 1, 2, 4, 8, 12 and 16 weeks post-dose
  To characterize the PK of AZD2693 following SC administration of SAD of AZD2693
Time to reach maximum observed concentration following drug administration (tmax) | At Day 1 pre-dose, 0.25h, 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 5h, 6h, 8h, 12h, 24h, 36h, 48h and 72h post-dose and 1, 2, 4, 8, 12 and 16 weeks post-dose
  To characterize the PK of AZD2693 following SC administration of SAD of AZD2693
Apparent terminal elimination half-life associated with the terminal slope (λz) of the semi-logarithmic concentration-time curve, estimated as (ln2)/λz (t½λz) | At Day 1 pre-dose, 0.25h, 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 5h, 6h, 8h, 12h, 24h, 36h, 48h and 72h post-dose and 1, 2, 4, 8, 12 and 16 weeks post-dose
  To characterize the PK of AZD2693 following SC administration of SAD of AZD2693.
Apparent total body clearance of drug from plasma after extravascular administration calculated as Dose/AUC (CL/F) | At Day 1 pre-dose, 0.25h, 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 5h, 6h, 8h, 12h, 24h, 36h, 48h and 72h post-dose and 1, 2, 4, 8, 12 and 16 weeks post-dose
  To characterize the PK of AZD2693 following SC administration of SAD of AZD2693
Apparent volume of distribution for parent drug at terminal phase (extravascular administration), estimated by dividing CL/F by λz (Vz/F) | At Day 1 pre-dose, 0.25h, 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 5h, 6h, 8h, 12h, 24h, 36h, 48h and 72h post-dose and 1, 2, 4, 8, 12 and 16 weeks post-dose
  To characterize the PK of AZD2693 following SC administration of SAD of AZD2693
Mean residence time (MRT) | At Day 1 pre-dose, 0.25h, 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 5h, 6h, 8h, 12h, 24h, 36h, 48h and 72h post-dose and 1, 2, 4, 8, 12 and 16 weeks post-dose
  To characterize the PK of AZD2693 following SC administration of SAD of AZD2693
Terminal elimination rate constant, estimated by log-linear least-squares regression of the terminal part of the concentration-time curve (λz) | At Day 1 pre-dose, 0.25h, 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 5h, 6h, 8h, 12h, 24h, 36h, 48h and 72h post-dose and 1, 2, 4, 8, 12 and 16 weeks post-dose
  To characterize the PK of AZD2693 following SC administration of SAD of AZD2693
Time delay between drug administration and the first observed concentration in plasma (tlag) | At Day 1 pre-dose, 0.25h, 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 5h, 6h, 8h, 12h, 24h, 36h, 48h and 72h post-dose and 1, 2, 4, 8, 12 and 16 weeks post-dose
  To characterize the PK of AZD2693 following SC administration of SAD of AZD2693
Time of the last quantifiable concentration (tlast) | At Day 1 pre-dose, 0.25h, 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 5h, 6h, 8h, 12h, 24h, 36h, 48h and 72h post-dose and 1, 2, 4, 8, 12 and 16 weeks post-dose
  To characterize the PK of AZD2693 following SC administration of SAD of AZD2693
Cumulative fraction (%) of dose excreted unchanged into the urine from time zero to the last measured time point [fe(0-last)] | At Day 1 pre-dose, 0-6h, 6-12h and then 0-12h intervals up to 72h post-dose
  To characterize the PK of AZD2693 following SC administration of SAD of AZD2693
Cumulative amount of analyte excreted into the urine from time zero through the last sampling interval [Ae(0-last)] | At Day 1 pre-dose, 0-6h, 6-12h and then 0-12h intervals up to 72h post-dose
  To characterize the PK of AZD2693 following SC administration of SAD of AZD2693
Renal clearance of drug from plasma, estimated by dividing Ae(0-t) by AUC(0-t) where the 0-t interval is the same for both Ae and AUC [CLR] | At Day 1 pre-dose, 0-6h, 6-12h and then 0-12h intervals up to 72h post-dose
  To characterize the PK of AZD2693 following SC administration of SAD of AZD2693
Amount of analyte excreted into the urine from time t1 to t2 [Ae(t1-t2)] | At Day 1 pre-dose, 0-6h, 6-12h and then 0-12h intervals up to 72h post-dose
  To characterize the PK of AZD2693 following SC administration of SAD of AZD2693
Fraction of dose excreted unchanged into the urine from time t1 to t2 [fe(t1-t2)] | At Day 1 pre-dose, 0-6h, 6-12h and then 0-12h intervals up to 72h post-dose
  To characterize the PK of AZD2693 following SC administration of SAD of AZD2693

CONTACTS AND LOCATIONS:
Overall Officials: David Han, MD, Principal Investigator — Parexel Early Clinical Unit - Los Angeles
Locations (1):
- Research Site, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Armisen J, Rauschecker M, Sarv J, Liljeblad M, Wernevik L, Niazi M, Knochel J, Eklund O, Sandell T, Sherwood J, Bergenholm L, Hallen S, Wang S, Kamble P, Bhat M, Maxvall I, Wang Y, Lee RG, Bhanot S, Guo S, Romeo S, Lawitz E, Fjellstrom O, Linden D, Blau JE, Loomba R. AZD2693, a PNPLA3 antisense oligonucleotide, for the treatment of MASH in 148M homozygous participants: Two randomized phase I trials. J Hepatol. 2025 Jul;83(1):31-42. doi: 10.1016/j.jhep.2024.12.046. Epub 2025 Jan 9. PMID 39798707